CLINICAL TRIAL: NCT00258076
Title: Open-Label, Randomized, Partially Balanced, Incomplete Block Design Sudy to Evaluate the Hormone Exposure From Commercial ORTHO EVRA�
Brief Title: A Study to Evaluate the Hormone Exposure From Multiple Commercial Lots of ORTHO EVRA (a Transdermal Contraceptive Patch)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR002215
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Contraception; Female Contraception
Keywords: Transdermal contraception; contraceptive; hormonal, steroid contraception; ethinyl estradiol; progesterone; EVRA

ARMS (1):
- 001 (Experimental): EVRA transdermal contraceptive patch 6 mg NGMN and 0.75 mg EE
  Interventions: Drug: EVRA transdermal contraceptive patch 6 mg NGMN and 0.75 mg EE

INTERVENTIONS:
Drug: EVRA transdermal contraceptive patch 6 mg NGMN and 0.75 mg EE

SUMMARY:
The objective of this study is to estimate the exposure to the hormones norelgestromin, norgestrel, and ethinyl estradiol in the bloodstream of healthy female volunteers across multiple commercial lots of ORTHO EVRAÂ® (a transdermal contraceptive patch) and to compare these data to historical hormonal exposure data from one ORTHO EVRAÂ® clinical development lot.

DETAILED DESCRIPTION:
This multicenter, open-label, randomized, partially-balanced, incomplete block design study will consist of a pre-treatment phase (a screening period lasting up to 21 days), an open-label treatment phase (three 7-day treatment periods separated by 21-day washouts), and a post-treatment phase (a follow-up or early withdrawal visit). Total participation in the study is approximately 67 days. Approximately 52 subjects will be enrolled. The study population comprises healthy women, ages 18 to 45 years inclusive, who weigh at least 110 pounds, have a body mass index (BMI) between 16 and 29.9 kg per meter squared.

An ORTHO EVRA® patch from 1 of the 13 selected commercial lots will be applied to the buttock of each subject and worn for 7 days. Patches will be applied on Days 1, 29, and 57 by the investigator or designated study unit personnel. Each patch will be worn on the upper outer quadrant of the same buttock, but the 3 patches will not necessarily be placed in the exact same position. The investigator or designated study unit personnel will remove the patches on Days 8, 36, and 64 and will evaluate the adhesion of the patches before removal.

Subjects will be confined to the study unit for blood sample collections for determination of NGMN, NG, and EE serum concentrations. Blood samples will be collected (via venipuncture) immediately before and at specified time points after each patch application. Pharmacokinetic parameters of NGMN, NG, and EE, including Cmax, tmax, and AUC for each treatment will be estimated by standard methods. Safety will be assessed throughout the study, and will be based on adverse events and changes in physical and gynecologic examinations (including breast examinations), vital signs, electrocardiograms (ECGs), and clinical laboratory test results. Three 7-day treatment periods, separated by 21-day washouts, as follows: Each ORTHO EVRA® patch will be worn on the buttock (upper outer quadrant) for 7 days. Twenty one days after completing each treatment, subjects will cross over to the next treatment for 7 days. The patch will be applied to the upper outer quadrant of the same buttock as before, but not necessarily in the exact same spot.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are not pregnant (as demonstrated by negative pregnancy tests at screening and before admission for each treatment period) and who have completed their last term pregnancy at least 60 days before the admission visit
* confirmed to be in good health as determined by medical history, physical examination (including vital signs), gynecologic examination (including breast examination), and laboratory test results
* have a history of regular menstrual cycles, weigh at least 110 pounds (50 kilograms), have a body mass index (BMI) between 16 and 29.9 kg per meter squared, a hematocrit of at least 36% at screening, and a ferritin level above the lower limit of normal
* are nonsmokers and have not used any tobacco products for at least 6 months before study admission
* agree not to use any prescription or nonprescription medications for the duration of the study, and if the subject or her male partner are not surgically sterile, agree to continue to use a non-hormone-containing intrauterine device (IUD) or one of the following methods of double-barrier contraception during participation in the study: condoms and foam, diaphragm and gel, or cervical cap and gel.

Exclusion Criteria:

* Subjects with a history or presence of disorders commonly accepted as contraindications to sex hormonal therapy including, but not limited to: deep vein thrombophlebitis or thromboembolic disorders, cerebral vascular or coronary artery disease, chronic untreated hypertension or migraines, benign or malignant liver tumor which developed during the use of oral contraceptives or other estrogen-containing products, or known or suspected estrogen-dependent neoplasia
* presence of disorders commonly accepted as contraindications to combined oral contraceptive therapy including, but not limited to: undiagnosed abnormal vaginal bleeding, any neurovascular lesion of the eye or serious visual disturbance, any impairment of liver function, liver disease, or kidney disease
* currently pregnant or breast feeding, or have evidence of cervical dysplasia (as documented by a Pap smear within 6 months before randomization)
* has used steroid hormonal therapy within 30 days before the first admission visit, received a Depo Provera® injection within 6 months of the first admission visit, received a Lunelle® injection within 60 days before the first admission visit, currently has Norplant® in place, or has had removal of Norplant within the 60 days before the first admission visit, or has used a steroid hormone-containing intrauterine device (IUD) within 3 months of randomization
* has elevated blood pressure (sitting systolic BP >140 mm Hg and/or diastolic BP >90 mm Hg)
* has a history or presence of hypersensitivity in response to topical applications (bandages, surgical tape, etc.) or has active inflammation of the skin (dermatitis) or other skin conditions (dermatosis).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2004-04; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
A comparison of the exposure and pharmacokinetics of NGMN, NG, and EE after a single patch application of different commercial lots of ORTHO EVRA and a comparison of these data to historical hormonal data from a clinical development patch.

SECONDARY OUTCOMES:
An assessment of safety from screening to final visit (incidence of adverse events, changes in physical, gynecologic and breast examinations, vital signs, laboratory tests and electrocardiogram results).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Open-Label, Randomized, Partially Balanced, Incomplete Block Design Study to Evaluate the Hormone Exposure From Commercial ORTHO EVRA� — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=459&filename=CR002215_CSR.pdf